CLINICAL TRIAL: NCT01870856
Title: Evaluation of Lid Wiper Epitheliopathy With and Without Daily Disposable Contact Lenses
Brief Title: Lid Wiper Epitheliopathy Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary efficacy was not demonstrated in Stage 1
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-13-005
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Lid Wiper Epitheliopathy
Keywords: Ocular discomfort; Contact lenses; Myopia
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Spectacles, Stage 1 (Experimental): Spectacles per participant's habitual perscription worn for 2 weeks
  Interventions: Device: Spectacles
- 1-DAY ACUVUE, Stage 1 (Active Comparator): Etafilcon A contact lenses worn in both eyes at least 5 days per week, at least 6 hours per day, for 2 weeks in a daily disposable mode
  Interventions: Device: Etafilcon A contact lenses
- DAILIES TOTAL1, Stage 2 (Experimental): Delefilcon A contact lenses worn in both eyes at least 5 days per week, at least 6 hours per day, for 2 weeks in a daily disposable mode
  Interventions: Device: Delefilcon A contact lenses
- 1-DAY ACUVUE, Stage 2 (Active Comparator): Etafilcon A contact lenses worn in both eyes at least 5 days per week, at least 6 hours per day, for 2 weeks in a daily disposable mode
  Interventions: Device: Etafilcon A contact lenses

INTERVENTIONS:
Device: Spectacles — Per participant's habitual prescription
  Arms: Spectacles, Stage 1
Device: Delefilcon A contact lenses — Silicone hydrogel single vision contact lenses
  Other Names: DAILIES TOTAL1®
  Arms: DAILIES TOTAL1, Stage 2
Device: Etafilcon A contact lenses — Hydrogel single vision contact lenses
  Other Names: 1-DAY ACUVUE®
  Arms: 1-DAY ACUVUE, Stage 1; 1-DAY ACUVUE, Stage 2

SUMMARY:
The purpose of this study is to evaluate the effect of contact lens lubricity on lid wiper epitheliopathy (LWE) in symptomatic contact lens wearers. LWE is defined as an alteration of that portion of the marginal conjunctival epithelium of the upper eyelid that wipes the ocular surface during blinking.

DETAILED DESCRIPTION:
This study will be conducted in two stages. In Stage 1, participants will wear either spectacles or contact lenses for two weeks to determine the impact of interruption of contact lens wear on LWE. In Stage 2, a second cohort of participants will wear one of two contact lens brands for two weeks, and LWE and ocular discomfort will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document.
* Severe lid wiper epitheliopathy (upper lid) in either eye.
* Currently wearing spherical daily disposable soft contact lenses or daily wear soft contact lenses in both eyes with at least 3 months of contact lens wearing experience.
* Symptomatic as determined by the SPEED questionnaire.
* Willing to follow visit schedule.
* Habitual contact lens power with the range of -1.00 to -6.00 diopters (D) with best corrected distance visual acuity greater than or equal to 20/25 in each eye.
* Astigmatism less than or equal to 0.75D.
* Possess spectacles which provide visual acuity of at least 20/25 in each eye.
* Willing and able to complete daily diaries.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury within 12 weeks immediately prior to enrollment.
* Any ocular condition that would contraindicate contact lens wear.
* Any use of systemic or ocular medications that would contraindicate contact lens wear, as determined by the investigator.
* Currently wearing toric or multifocal soft contact lenses.
* Participation in a clinical study (including contact lens or contact lens care product) within the previous 30 days.
* Routinely sleeps in lenses for at least 1 night per week.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Brobst, OD, FAAO, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 23 study centers located in the US.
Pre-assignment Details: Of the 187 enrolled, 135 participants were exited as screen failures prior to randomization. This reporting group includes all randomized participants. Results from Stage 1 were planned to be used to appropriately power Stage 2 of the study. Since primary efficacy cannot be demonstrated in Stage 1, Stage 2 of this study was not conducted.
Groups:
- 1-DAY ACUVUE, Stage 1: Contact lenses worn bilaterally (in both eyes) at least 5 days per week, at least 6 hours per day, for 2 weeks in a daily disposable mode
Period: Overall Study
Arm/Group | Spectacles, Stage 1 | 1-DAY ACUVUE, Stage 1
Started | 25 | 27
Completed | 25 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants/eyes exposed to investigational products (test and control).
Groups:
- Total: Total of all reporting groups
Arm/Group | Spectacles, Stage 1 | 1-DAY ACUVUE, Stage 1 | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.9) | 34.1 (9.4) | 34.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Percent of Eyes Experiencing at Least 1 Grade Reduction in LWE at 2 Weeks
Description: LWE was measured by slit lamp evaluation of fluorescein and lissamine green staining of the upper eyelid. LWE was graded on a scale from 0 to 3, where 0=none and 3=severe. The percent of eyes experiencing at least a 1 grade reduction in LWE (from baseline) at the 2-week visit was compared between groups. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 2
Population: This analysis population includes all randomized subjects who did not meet the critical deviation criteria as specified in the Deviations and Evaluability Plan. Denominator for percentages is the number of subjects with data available at both time points.
Measure: Number; unit: percentage of subjects
Arm/Group | Spectacles, Stage 1 | 1-DAY ACUVUE, Stage 1
Number analyzed (Participants) | 21 | 21
percentage of subjects | 100 | 81

2. Primary Outcome: Stage 2: Percent of Eyes Experiencing at Least 1 Grade Reduction in LWE at 2 Weeks
Description: This outcome measure was not evaluated since primary efficacy was not demonstrated.
Time Frame: Baseline, Week 2
Groups:
- DAILIES TOTAL 1, Stage 2; 1-DAY ACUVUE, Stage 2: Contact lenses worn bilaterally (in both eyes) at least 5 days per week, at least 6 hours per day, for 2 weeks in a daily disposable mode
Arm/Group | DAILIES TOTAL 1, Stage 2 | 1-DAY ACUVUE, Stage 2
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Stage 2: Change From Baseline in Ocular Discomfort Score (as Measured by SPEED) at 2 Weeks
Description: This outcome measure was not evaluated since primary efficacy was not demonstrated.
Time Frame: Baseline, Week 2
Arm/Group | DAILIES TOTAL 1, Stage 2 | 1-DAY ACUVUE, Stage 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from 15 Jul 2013 to 29 Oct 2013. Reports of AEs were obtained through spontaneous comments from the subjects and through observations by the Investigator as outlined in the study protocol.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or clinical signs in subjects, users or other persons, whether or not related to the investigational device (test article). This analysis group includes all subjects/eyes exposed to investigational products (test and control).
Arm/Group | Spectacles, Stage 1 | 1-DAY ACUVUE, Stage 1
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.